CLINICAL TRIAL: NCT03911674
Title: Effects of Oral Stimulation on Feeding Performance, Length of Hospital Stay and Anthropometric Variables of Preterm Infants
Brief Title: Effects of Oral Stimulation in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEU-0013
Record Dates: First submitted 2019-03-31; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Premature Infant; Eating Disorder
MeSH Terms: conditions — Premature Birth; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral stimulation (Experimental): Oral stimulation protocol: manual stimulation of the oral sucking
  Interventions: Other: Oral manual stimulation of feeding in preterm infants
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Oral manual stimulation of feeding in preterm infants — Manual stimulation of the cheeks (internal and external), lips, gums, tongue and palate by finger-strokin.
  Arms: Oral stimulation

SUMMARY:
Preterm infants with gestational age inferior to 34 weeks were included in the study. A prospective experimental group received the oral stimulation protocol and the effects of the intervention were compared with a historical control group that did not receive any oral stimulation intervention.

The study hypothesis is that oral stimulation in preterm infants has beneficial effects on the feeding performance, the length of hospitalization and anthropometric variables, including weight at discharge, height at discharge and head circumference at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age inferior to 34 weeks

Exclusion Criteria:

* Instability caused by respiratory, cardiac or gastrointestinal issues
* Orofacial malformations.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Gestational age at the initiation of oral feeding | Up to 46 weeks
Weight at discharge (g) | Up to 46 weeks
Height at discharge (cm) | Up to 46 weeks
Head circumference at discharge (cm) | Up to 46 weeks
Days of enteral nutrition | Up to 46 weeks
Gestational age at discharge (weeks) | Up to 46 weeks
Total length of hospitalization | Up to 46 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CEU San Pablo University, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No